CLINICAL TRIAL: NCT05603702
Title: STTEPP: Safety, Tolerability and Dose Limiting Toxicity of Lacosamide in Patients With Painful Chronic Pancreatitis
Acronym: STTEPP
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Evan Fogel, Stuart Sherman Professor in Gastroenterology & Hepatology, Lehman, Bucksot and Sherman Section of Pancreatobiliary Endoscopy Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHHBRBAPSM35; 1R01DK132709-01 (NIH)
Record Dates: First submitted 2022-10-18; First posted 2022-11-03 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Chronic Pain Syndrome; Chronic Pancreatitis; Hyperalgesia; Opioid Use Disorder; Opioid-Related Disorders; Opioid Dependence; Chronic Abdominal Pain; ERCP; Pancreatic Surgery
Keywords: Pancreatitis; Pancreatitis, chronic; Chronic pain; Pain; Pancreatic Diseases; Digestive System Diseases
MeSH Terms: conditions — Chronic Pain; Pancreatitis, Chronic; Hyperalgesia; Opioid-Related Disorders; Pancreatitis; Pain; Pancreatic Diseases; Digestive System Diseases | interventions — Lacosamide

STUDY DESIGN:
Intervention Model Description: 1. Patients in the first cohort are treated at dose level 1.
  2. Once a cohort of three patients has been recruited at a given dose level, recruitment will temporarily be held until all three patients have been evaluated for delayed adverse events, at 21 ±3 days following completion of drug therapy.
  3. To assign a dose to the next cohort of patients, conduct dose escalation/de-escalation according to BOIN design rules.
  4. Repeat step 2 until the maximum sample size of 24 is reached or stop the trial if the number of patients treated at the current dose reaches 15.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation Level (Experimental): In the first 3-patient cohort, the dose of lacosamide given is 50mg/d BID. Enrollment to the next higher dose cohort will be initiated only if none of the 3 participants exhibits a DLT in the 21 ±3 days following completion of the 7 day drug therapy. Dose escalation will proceed according to the Bayesian optimal interval (BOIN) design at incremental increase of 100mg/day in two divided doses. The maximum daily dose of lacosamide will be 400mg/day.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Study Visit 1: Baseline study assessments will be made and questionnaires completed in person, on day 0. Drug treatment days will then occur on days 1-7. Study Visit 2: Following completion of the 7-day drug treatment period, participants will have a face-to-face clinic visit on day 8 (with a 3 day grace period), where similar assessments and questionnaires will again be completed. Participants will return all unused drug at this visit, for disposal and to monitor compliance. A follow-up phone visit will occur on day 21 (with a 3 day window) to assess for adverse events and medication changes
  Other Names: VIMPAT

SUMMARY:
The investigators propose to conduct a dose-escalation trial of an FDA-approved antiepileptic drug, lacosamide, added to opioid therapy in patients with chronic abdominal pain from chronic pancreatitis (CP). This pilot trial will test the feasibility of the study design and provide reassurance regarding the tolerability and safety of lacosamide used concomitantly with opioids in this patient population to reduce the condition known clinically as opioid-induced hyperalgesia (OIH).

DETAILED DESCRIPTION:
One rather pronounced adverse off-target effect of opioids is an increasing sensitivity to noxious stimuli, even evolving a painful response to previously non-noxious stimuli, known clinically as opioid-induced hyperalgesia (OIH). Based on pre-clinical published data, therapeutic targeting of the sodium channel NaV1.7 may address one of the mechanisms that limits opioid efficacy for controlling pain. The investigators hypothesize that lacosamide, an FDA-approved antiepileptic drug that targets NaV1.7, used concomitantly with opioids will improve the opioid efficacy for controlling pain in patients with chronic pancreatitis (CP). However, there are no preliminary data available evaluating lacosamide in this patient population. Therefore, a phase 1 trial is necessary.

The investigators will employ the Bayesian optimal interval (BOIN) design to find the Maximum Tolerated Dose (MTD). The investigators will enroll and treat patients in cohorts of size 3. The initial dose will be 50mg po bid (100mg/day), followed by incremental increases of 100mg/day in two divided doses. The maximum daily dose of lacosamide will be 400mg/day. Duration of lacosamide administration will be 7 days at each dose level. Follow-up laboratory parameters (as obtained at study entry) will be obtained on day 8 (with a 3 day window) after therapy is completed. A follow-up phone visit will occur on day 21 (with a 3-day window) to assess for adverse events and medication changes.

It is anticipated that lacosamide will prove to be safe and well-tolerated. The results of this pilot study will then support proceeding with a subsequent phase 2 trial assessing the efficacy of lacosamide added to opioid therapy to alleviate abdominal pain from CP. The investigators further anticipate that lacosamide combined with opiates will substantially lower the opioid dose necessary for adequate pain relief and serve to substantially improve the safety profile of opioid use for CP.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent and HIPAA authorization for release of personal health information;
2. ≥ 18 years old at the time of informed consent;
3. suspected (YELLOW 2 or 3) or definite diagnosis of CP, as per CPDPC PROCEED study definition with ongoing symptoms of abdominal pain;
4. patients must be maintained on an opioid (except methadone or suboxone) for 4 weeks prior to enrollment for treatment of abdominal pain related to pancreatitis;
5. ongoing symptoms of abdominal pain even with opioid use (VAS and BPI average score ≥4, at enrollment);
6. ECOG Performance Status of 0-2;(Oken et al., 1982)
7. ability to swallow and tolerate oral tablets;
8. females of childbearing potential must have a negative pregnancy test;
9. the following laboratory parameters must be met: WBC count ≥ 3.0 K/mm3, absolute neutrophil count ≥ 1.5 K/mm3, hemoglobin ≥ 9 g/dL, platelets ≥ 75 K/mm3, creatinine ≤ 1.5 mg/dl, bilirubin ≤ 1.5 x ULN, AST ≤ 3 x ULN, ALT ≤ 3 x ULN; normal PR interval on baseline 12-lead EKG.

Exclusion Criteria:

1. subjects with indeterminate CP (YELLOW 1) as per PROCEED criteria;
2. treatment with any investigational agent within 30 days prior to registration, or concurrent participation in a clinical trial which involves another investigational agent;
3. rapidly escalating pain that requires parenteral (intravenous or intramuscular) opioid therapy within 30 days of enrollment;
4. known hypersensitivity/allergic reaction to lacosamide, carbamazepine or oxcarbazepine;
5. pregnant or breastfeeding;
6. patient who has a diagnosis of epilepsy and/or is currently taking anti-epileptic drugs (other than gabapentin and pregabalin);
7. abdominal surgery or pain intervention (ERCP with sphincterotomy/stent/stone removal; celiac plexus block) within 90 days of enrollment.
8. hospitalization for pancreatitis exacerbation or pain management within 30 days of enrollment
9. patient who currently takes Suboxone or Methadone.
10. other factors which might explain the patient's ongoing symptoms, at the discretion of the enrolling physician.
11. history of autoimmune or traumatic pancreatitis, or sentinel attack of acute necrotizing pancreatitis which results in suspected disconnected duct syndrome.
12. primary pancreatic tumors- pancreatic ductal adenocarcinoma, suspected cystic neoplasm (>1cms in size or main duct involvement), neuroendocrine tumors, and other uncommon tumors.
13. pancreatic metastasis from other malignancies.
14. history of solid organ transplant, HIV/AIDS.
15. known isolated pancreatic exocrine insufficiency (e.g. in the absence of any eligible inclusion criteria).
16. participants must not have medical or psychiatric illnesses or ongoing substance abuse that in the investigator's opinion would compromise their ability to tolerate study interventions or participate in follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity of lacosamide in combination with opioids in CP patients will be measured by the number of grade 3 or4 toxicities reported via the CTCAE v5.0, between Day 1 through 21 day follow up. | Day 1, 21 day follow up
  Dose-limiting toxicity of combination lacosamide and opioids. Patients will be examined and graded for subjective/objective evidence of developing grade 3 or 4 toxicities according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Tolerability of lacosamide in combination with opioids in CP patients will be evaluated by the percentage of compliance in taking lacosamide pills as directed between Day 1 and Day 7. | Day 1, Day 7
  Tolerability will be assessed by compliance with the intervention. Subjects will be evaluated for completing the 7-day trial. The percent of subjects taking 100%, 75%, 50% and <50% of tablets will be recorded.
Feasibility of performance of a pilot study adding lacosamide to opioid therapy in CP patients based on recruitment rate: measured by the proportion of eligible patients who continue from the screening visit to the enrollment visit. | Screening visit, Enrollment visit
  Recruitment rate (proportion of eligible patients approached who agree to participate)
Feasibility of performance of a pilot study adding lacosamide to opioid therapy in CP patients based on retention rate measured by the change from the screening visit to the 21 day follow-up visit. | Screening visit, 21 day follow-up
  Dropout rate, including qualitative assessment of barriers to retention.

SECONDARY OUTCOMES:
Efficacy of adding lacosamide to opioid therapy for the treatment of abdominal pain due to CP by a 50% decrease in the VAS score from the Screening visit to the Follow-up visit day 8.. | Screening visit, Day 8
  Visual Analog Score (VAS) - a 50% decrease in score from Screening visit to Follow-up visit day 8.
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Efficacy of adding lacosamide to opioid therapy for the treatment of abdominal pain due to CP by a 50% decrease in BPI-SF average pain score from the Screening visit to the Day 8 visit. | Screening visit, Day 8
  Brief Pain Inventory (BPI), short form average score - a 50% decrease in total score from Screening visit to Follow-up visit day 8 The BPI-SF is a validated self-reported tool that evaluates pain severity and pain interference with daily activities at the time of assessment. Possible scores for pain severity range from 0 to 10 (higher scores reflect more severe pain)
Efficacy of adding lacosamide to opioid therapy for the treatment of abdominal pain due to CP by a 50% decrease in total score of the Compat-SF pain severity from the Screening visit to Follow-up visit day 8. | Screening visit, Day 8
  Compat-SF total score - a 50% decrease in total score from Screening visit to Follow-up visit day 8 The COMPAT-SF is a validated self-reported tool specifically designed for patients with pancreatic disease. Scores for pain severity (average, worst, and least) range from 0 to 10 (higher corresponds to more pain); scores for pain triggers (including food, exercise, and thermal changes) are scored on a scale from never to always (never, rarely, sometimes, very often, always); scores for pain symptom characteristics (cramping, shooting, stabbing) are scored on a scale from 0 (none) to 10 (worst possible).
Efficacy of adding lacosamide to opioid therapy for the treatment of abdominal pain due to CP by a 25% decrease in morphine milligram equivalents (MME) of opioid use from the Screening visit to Follow-up visit day 8. | Screening visit, Day 8
  Opioid use will decrease by 25% from screening visit to Follow-up visit day 8. Patients will be asked to track all opioids taken on a drug diary from the screening visit through day 8 of study intervention. MME will be calculated to compare level of MME from screening visit to day 8.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Unalp-Arida, MD, PhD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient data may be shared with investigators from outside institutions for ancillary studies upon request. Requests should be made to study principal investigator at efogel@iu.edu.
Time Frame: Data will be available at the close of the study and for 5 years subsequent.
Access Criteria: Individual requests for data sharing can be made to: efogel@iu.edu

REFERENCES:
- [Result] Agarwal D, Udoji MA, Trescot A. Genetic Testing for Opioid Pain Management: A Primer. Pain Ther. 2017 Jun;6(1):93-105. doi: 10.1007/s40122-017-0069-2. Epub 2017 Apr 13. PMID 28409480
- [Result] Angst MS, Clark JD. Opioid-induced hyperalgesia: a qualitative systematic review. Anesthesiology. 2006 Mar;104(3):570-87. doi: 10.1097/00000542-200603000-00025. PMID 16508405
- [Result] Bannister K. Opioid-induced hyperalgesia: where are we now? Curr Opin Support Palliat Care. 2015 Jun;9(2):116-21. doi: 10.1097/SPC.0000000000000137. PMID 25872113
- [Result] Bannister K, Bee LA, Dickenson AH. Preclinical and early clinical investigations related to monoaminergic pain modulation. Neurotherapeutics. 2009 Oct;6(4):703-12. doi: 10.1016/j.nurt.2009.07.009. PMID 19789074
- [Result] Ben-Menachem E, Biton V, Jatuzis D, Abou-Khalil B, Doty P, Rudd GD. Efficacy and safety of oral lacosamide as adjunctive therapy in adults with partial-onset seizures. Epilepsia. 2007 Jul;48(7):1308-17. doi: 10.1111/j.1528-1167.2007.01188.x. PMID 17635557
- [Result] Cawello W. Clinical pharmacokinetic and pharmacodynamic profile of lacosamide. Clin Pharmacokinet. 2015 Sep;54(9):901-14. doi: 10.1007/s40262-015-0276-0. PMID 25957198
- [Result] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Result] Colvin LA, Fallon MT. Opioid-induced hyperalgesia: a clinical challenge. Br J Anaesth. 2010 Feb;104(2):125-7. doi: 10.1093/bja/aep392. No abstract available. PMID 20086062
- [Result] Cote GA, Yadav D, Slivka A, Hawes RH, Anderson MA, Burton FR, Brand RE, Banks PA, Lewis MD, Disario JA, Gardner TB, Gelrud A, Amann ST, Baillie J, Money ME, O'Connell M, Whitcomb DC, Sherman S; North American Pancreatitis Study Group. Alcohol and smoking as risk factors in an epidemiology study of patients with chronic pancreatitis. Clin Gastroenterol Hepatol. 2011 Mar;9(3):266-73; quiz e27. doi: 10.1016/j.cgh.2010.10.015. Epub 2010 Oct 26. PMID 21029787
- [Result] Cote GA, Durkalski-Mauldin VL, Serrano J, Klintworth E, Williams AW, Cruz-Monserrate Z, Arain M, Buxbaum JL, Conwell DL, Fogel EL, Freeman ML, Gardner TB, van Geenen E, Groce JR, Jonnalagadda SS, Keswani RN, Menon S, Moffatt DC, Papachristou GI, Ross A, Tarnasky PR, Wang AY, Wilcox CM, Hamilton F, Yadav D; SHARP Consortium. SpHincterotomy for Acute Recurrent Pancreatitis Randomized Trial: Rationale, Methodology, and Potential Implications. Pancreas. 2019 Sep;48(8):1061-1067. doi: 10.1097/MPA.0000000000001370. PMID 31404020
- [Result] Cotton PB, Durkalski V, Romagnuolo J, Pauls Q, Fogel E, Tarnasky P, Aliperti G, Freeman M, Kozarek R, Jamidar P, Wilcox M, Serrano J, Brawman-Mintzer O, Elta G, Mauldin P, Thornhill A, Hawes R, Wood-Williams A, Orrell K, Drossman D, Robuck P. Effect of endoscopic sphincterotomy for suspected sphincter of Oddi dysfunction on pain-related disability following cholecystectomy: the EPISOD randomized clinical trial. JAMA. 2014 May;311(20):2101-9. doi: 10.1001/jama.2014.5220. PMID 24867013
- [Result] Dean L. Lacosamide Therapy and CYP2C19 Genotype. 2018 Apr 18. In: Pratt VM, Scott SA, Pirmohamed M, Esquivel B, Kattman BL, Malheiro AJ, editors. Medical Genetics Summaries [Internet]. Bethesda (MD): National Center for Biotechnology Information (US); 2012-. Available from http://www.ncbi.nlm.nih.gov/books/NBK493589/ PMID 29671994
- [Result] Deuis JR, Dekan Z, Wingerd JS, Smith JJ, Munasinghe NR, Bhola RF, Imlach WL, Herzig V, Armstrong DA, Rosengren KJ, Bosmans F, Waxman SG, Dib-Hajj SD, Escoubas P, Minett MS, Christie MJ, King GF, Alewood PF, Lewis RJ, Wood JN, Vetter I. Pharmacological characterisation of the highly NaV1.7 selective spider venom peptide Pn3a. Sci Rep. 2017 Jan 20;7:40883. doi: 10.1038/srep40883. PMID 28106092
- [Result] Due MR, Piekarz AD, Wilson N, Feldman P, Ripsch MS, Chavez S, Yin H, Khanna R, White FA. Neuroexcitatory effects of morphine-3-glucuronide are dependent on Toll-like receptor 4 signaling. J Neuroinflammation. 2012 Aug 16;9:200. doi: 10.1186/1742-2094-9-200. PMID 22898544
- [Result] Due MR, Yang XF, Allette YM, Randolph AL, Ripsch MS, Wilson SM, Dustrude ET, Khanna R, White FA. Carbamazepine potentiates the effectiveness of morphine in a rodent model of neuropathic pain. PLoS One. 2014 Sep 15;9(9):e107399. doi: 10.1371/journal.pone.0107399. eCollection 2014. PMID 25221944
- [Result] Elmunzer BJ, Scheiman JM, Lehman GA, Chak A, Mosler P, Higgins PD, Hayward RA, Romagnuolo J, Elta GH, Sherman S, Waljee AK, Repaka A, Atkinson MR, Cote GA, Kwon RS, McHenry L, Piraka CR, Wamsteker EJ, Watkins JL, Korsnes SJ, Schmidt SE, Turner SM, Nicholson S, Fogel EL; U.S. Cooperative for Outcomes Research in Endoscopy (USCORE). A randomized trial of rectal indomethacin to prevent post-ERCP pancreatitis. N Engl J Med. 2012 Apr 12;366(15):1414-22. doi: 10.1056/NEJMoa1111103. PMID 22494121
- [Result] Fogel EL, Lehman GA, Tarnasky P, Cote GA, Schmidt SE, Waljee AK, Higgins PDR, Watkins JL, Sherman S, Kwon RSY, Elta GH, Easler JJ, Pleskow DK, Scheiman JM, El Hajj II, Guda NM, Gromski MA, McHenry L Jr, Arol S, Korsnes S, Suarez AL, Spitzer R, Miller M, Hofbauer M, Elmunzer BJ; US Cooperative for Outcomes Research in Endoscopy (USCORE). Rectal indometacin dose escalation for prevention of pancreatitis after endoscopic retrograde cholangiopancreatography in high-risk patients: a double-blind, randomised controlled trial. Lancet Gastroenterol Hepatol. 2020 Feb;5(2):132-141. doi: 10.1016/S2468-1253(19)30337-1. Epub 2019 Nov 25. PMID 31780277
- [Result] Gilron I, Bailey JM, Tu D, Holden RR, Weaver DF, Houlden RL. Morphine, gabapentin, or their combination for neuropathic pain. N Engl J Med. 2005 Mar 31;352(13):1324-34. doi: 10.1056/NEJMoa042580. PMID 15800228
- [Result] Goodman CW, Brett AS. Gabapentin and Pregabalin for Pain - Is Increased Prescribing a Cause for Concern? N Engl J Med. 2017 Aug 3;377(5):411-414. doi: 10.1056/NEJMp1704633. No abstract available. PMID 28767350
- [Result] Hall TC, Garcea G, Webb MA, Al-Leswas D, Metcalfe MS, Dennison AR. The socio-economic impact of chronic pancreatitis: a systematic review. J Eval Clin Pract. 2014 Jun;20(3):203-7. doi: 10.1111/jep.12117. Epub 2014 Mar 24. PMID 24661411
- [Result] Haugan F, Rygh LJ, Tjolsen A. Ketamine blocks enhancement of spinal long-term potentiation in chronic opioid treated rats. Acta Anaesthesiol Scand. 2008 May;52(5):681-7. doi: 10.1111/j.1399-6576.2008.01637.x. PMID 18419722
- [Result] Hearn L, Derry S, Moore RA. Lacosamide for neuropathic pain and fibromyalgia in adults. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD009318. doi: 10.1002/14651858.CD009318.pub2. PMID 22336864
- [Result] Hewitt DJ. The use of NMDA-receptor antagonists in the treatment of chronic pain. Clin J Pain. 2000 Jun;16(2 Suppl):S73-9. doi: 10.1097/00002508-200006001-00013. PMID 10870744
- [Result] Ibrahim SA, Albany Z, Albany C. Significant response to lacosamide in a patient with severe chemotherapy-induced peripheral neuropathy. J Community Support Oncol. 2015 May;13(5):202-4. doi: 10.12788/jcso.0136. PMID 26029937
- [Result] Isensee J, Krahe L, Moeller K, Pereira V, Sexton JE, Sun X, Emery E, Wood JN, Hucho T. Synergistic regulation of serotonin and opioid signaling contributes to pain insensitivity in Nav1.7 knockout mice. Sci Signal. 2017 Jan 10;10(461):eaah4874. doi: 10.1126/scisignal.aah4874. PMID 28074005
- [Result] Jo S, Bean BP. Lacosamide Inhibition of Nav1.7 Voltage-Gated Sodium Channels: Slow Binding to Fast-Inactivated States. Mol Pharmacol. 2017 Apr;91(4):277-286. doi: 10.1124/mol.116.106401. Epub 2017 Jan 24. PMID 28119481
- [Result] Li X, Angst MS, Clark JD. A murine model of opioid-induced hyperalgesia. Brain Res Mol Brain Res. 2001 Jan 31;86(1-2):56-62. doi: 10.1016/s0169-328x(00)00260-6. PMID 11165371
- [Result] Liang D, Shi X, Qiao Y, Angst MS, Yeomans DC, Clark JD. Chronic morphine administration enhances nociceptive sensitivity and local cytokine production after incision. Mol Pain. 2008 Feb 22;4:7. doi: 10.1186/1744-8069-4-7. PMID 18294378
- [Result] Minville V, Fourcade O, Girolami JP, Tack I. Opioid-induced hyperalgesia in a mice model of orthopaedic pain: preventive effect of ketamine. Br J Anaesth. 2010 Feb;104(2):231-8. doi: 10.1093/bja/aep363. Epub 2009 Dec 22. PMID 20031953
- [Result] Moore RA, Wiffen PJ, Derry S, McQuay HJ. Gabapentin for chronic neuropathic pain and fibromyalgia in adults. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD007938. doi: 10.1002/14651858.CD007938.pub2. PMID 21412914
- [Result] Mullady DK, Yadav D, Amann ST, O'Connell MR, Barmada MM, Elta GH, Scheiman JM, Wamsteker EJ, Chey WD, Korneffel ML, Weinman BM, Slivka A, Sherman S, Hawes RH, Brand RE, Burton FR, Lewis MD, Gardner TB, Gelrud A, DiSario J, Baillie J, Banks PA, Whitcomb DC, Anderson MA; NAPS2 Consortium. Type of pain, pain-associated complications, quality of life, disability and resource utilisation in chronic pancreatitis: a prospective cohort study. Gut. 2011 Jan;60(1):77-84. doi: 10.1136/gut.2010.213835. PMID 21148579
- [Result] Oken MM, Creech RH, Tormey DC, Horton J, Davis TE, McFadden ET, Carbone PP. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982 Dec;5(6):649-55. No abstract available. PMID 7165009
- [Result] Park KD, Yang XF, Dustrude ET, Wang Y, Ripsch MS, White FA, Khanna R, Kohn H. Chimeric agents derived from the functionalized amino acid, lacosamide, and the alpha-aminoamide, safinamide: evaluation of their inhibitory actions on voltage-gated sodium channels, and antiseizure and antinociception activities and comparison with lacosamide and safinamide. ACS Chem Neurosci. 2015 Feb 18;6(2):316-30. doi: 10.1021/cn5002182. Epub 2014 Dec 9. PMID 25418676
- [Result] Rao RD, Michalak JC, Sloan JA, Loprinzi CL, Soori GS, Nikcevich DA, Warner DO, Novotny P, Kutteh LA, Wong GY; North Central Cancer Treatment Group. Efficacy of gabapentin in the management of chemotherapy-induced peripheral neuropathy: a phase 3 randomized, double-blind, placebo-controlled, crossover trial (N00C3). Cancer. 2007 Nov 1;110(9):2110-8. doi: 10.1002/cncr.23008. PMID 17853395
- [Result] Rauck RL, Shaibani A, Biton V, Simpson J, Koch B. Lacosamide in painful diabetic peripheral neuropathy: a phase 2 double-blind placebo-controlled study. Clin J Pain. 2007 Feb;23(2):150-8. doi: 10.1097/01.ajp.0000210957.39621.b2. PMID 17237664
- [Result] Sarner M, Cotton PB. Classification of pancreatitis. Gut. 1984 Jul;25(7):756-9. doi: 10.1136/gut.25.7.756. PMID 6735257
- [Result] Serrano J, Andersen DK, Forsmark CE, Pandol SJ, Feng Z, Srivastava S, Rinaudo JAS; Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer: From Concept to Reality. Pancreas. 2018 Nov/Dec;47(10):1208-1212. doi: 10.1097/MPA.0000000000001167. PMID 30325859
- [Result] Shaibani A, Biton V, Rauck R, Koch B, Simpson J. Long-term oral lacosamide in painful diabetic neuropathy: a two-year open-label extension trial. Eur J Pain. 2009 May;13(5):458-63. doi: 10.1016/j.ejpain.2008.05.016. Epub 2008 Jul 10. PMID 18619874
- [Result] Shaibani A, Fares S, Selam JL, Arslanian A, Simpson J, Sen D, Bongardt S. Lacosamide in painful diabetic neuropathy: an 18-week double-blind placebo-controlled trial. J Pain. 2009 Aug;10(8):818-28. doi: 10.1016/j.jpain.2009.01.322. Epub 2009 May 5. PMID 19409861
- [Result] Sheets PL, Heers C, Stoehr T, Cummins TR. Differential block of sensory neuronal voltage-gated sodium channels by lacosamide [(2R)-2-(acetylamino)-N-benzyl-3-methoxypropanamide], lidocaine, and carbamazepine. J Pharmacol Exp Ther. 2008 Jul;326(1):89-99. doi: 10.1124/jpet.107.133413. Epub 2008 Mar 31. PMID 18378801
- [Result] Stohr T, Kupferberg HJ, Stables JP, Choi D, Harris RH, Kohn H, Walton N, White HS. Lacosamide, a novel anti-convulsant drug, shows efficacy with a wide safety margin in rodent models for epilepsy. Epilepsy Res. 2007 May;74(2-3):147-54. doi: 10.1016/j.eplepsyres.2007.03.004. Epub 2007 Apr 12. PMID 17433624
- [Result] Sutton KG, Martin DJ, Pinnock RD, Lee K, Scott RH. Gabapentin inhibits high-threshold calcium channel currents in cultured rat dorsal root ganglion neurones. Br J Pharmacol. 2002 Jan;135(1):257-65. doi: 10.1038/sj.bjp.0704439. PMID 11786502
- [Result] Tirkes T, Yadav D, Conwell DL, Territo PR, Zhao X, Venkatesh SK, Kolipaka A, Li L, Pisegna JR, Pandol SJ, Park WG, Topazian M, Serrano J, Fogel EL; Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer. Magnetic resonance imaging as a non-invasive method for the assessment of pancreatic fibrosis (MINIMAP): a comprehensive study design from the consortium for the study of chronic pancreatitis, diabetes, and pancreatic cancer. Abdom Radiol (NY). 2019 Aug;44(8):2809-2821. doi: 10.1007/s00261-019-02049-5. PMID 31089778
- [Result] Vardanyan A, Wang R, Vanderah TW, Ossipov MH, Lai J, Porreca F, King T. TRPV1 receptor in expression of opioid-induced hyperalgesia. J Pain. 2009 Mar;10(3):243-52. doi: 10.1016/j.jpain.2008.07.004. Epub 2008 Sep 6. PMID 18774343
- [Result] Venier J, Herrick R, Norris C, Liu S, Zhang L, Yuan Y Bayesian Optimal Interval (BOIN) Phase I Design (PID-862): Version 1.0.4. In. Houston, TX: The University of Texas MD Anderson Cancer Center.
- [Result] Vera-Portocarrero LP, Zhang ET, King T, Ossipov MH, Vanderah TW, Lai J, Porreca F. Spinal NK-1 receptor expressing neurons mediate opioid-induced hyperalgesia and antinociceptive tolerance via activation of descending pathways. Pain. 2007 May;129(1-2):35-45. doi: 10.1016/j.pain.2006.09.033. Epub 2006 Nov 22. PMID 17123731
- [Result] Wang Y, Wilson SM, Brittain JM, Ripsch MS, Salome C, Park KD, White FA, Khanna R, Kohn H. Merging Structural Motifs of Functionalized Amino Acids and alpha-Aminoamides Results in Novel Anticonvulsant Compounds with Significant Effects on Slow and Fast Inactivation of Voltage-gated Sodium Channels and in the Treatment of Neuropathic Pain. ACS Chem Neurosci. 2011 Jun 15;2(6):317-322. doi: 10.1021/cn200024z. PMID 21765969
- [Result] Wehler M, Reulbach U, Nichterlein R, Lange K, Fischer B, Farnbacher M, Hahn EG, Schneider T. Health-related quality of life in chronic pancreatitis: a psychometric assessment. Scand J Gastroenterol. 2003 Oct;38(10):1083-9. doi: 10.1080/00365520310005956. PMID 14621285
- [Result] Wiffen PJ, Derry S, Moore RA, McQuay HJ. Carbamazepine for acute and chronic pain in adults. Cochrane Database Syst Rev. 2011 Jan 19;(1):CD005451. doi: 10.1002/14651858.CD005451.pub2. PMID 21249671
- [Result] Wonder C (2016) Multiple cause of death data on CDC WONDER. In. Atlanta, GA US Department of Health and Human Services.
- [Result] Xie JY, Herman DS, Stiller CO, Gardell LR, Ossipov MH, Lai J, Porreca F, Vanderah TW. Cholecystokinin in the rostral ventromedial medulla mediates opioid-induced hyperalgesia and antinociceptive tolerance. J Neurosci. 2005 Jan 12;25(2):409-16. doi: 10.1523/JNEUROSCI.4054-04.2005. PMID 15647484
- [Result] Yadav D, Park WG, Fogel EL, Li L, Chari ST, Feng Z, Fisher WE, Forsmark CE, Jeon CY, Habtezion A, Hart PA, Hughes SJ, Othman MO, Rinaudo JAS, Pandol SJ, Tirkes T, Serrano J, Srivastava S, Van Den Eeden SK, Whitcomb DC, Topazian M, Conwell DL; Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer (CPDPC). PROspective Evaluation of Chronic Pancreatitis for EpidEmiologic and Translational StuDies: Rationale and Study Design for PROCEED From the Consortium for the Study of Chronic Pancreatitis, Diabetes, and Pancreatic Cancer. Pancreas. 2018 Nov/Dec;47(10):1229-1238. doi: 10.1097/MPA.0000000000001170. PMID 30325862
- [Result] Yang AL, Vadhavkar S, Singh G, Omary MB. Epidemiology of alcohol-related liver and pancreatic disease in the United States. Arch Intern Med. 2008 Mar 24;168(6):649-56. doi: 10.1001/archinte.168.6.649. PMID 18362258
- [Result] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Result] Yuan Y, Lin R, Li D, Nie L, Warren KE. Time-to-Event Bayesian Optimal Interval Design to Accelerate Phase I Trials. Clin Cancer Res. 2018 Oct 15;24(20):4921-4930. doi: 10.1158/1078-0432.CCR-18-0246. Epub 2018 May 16. PMID 29769209
- [Derived] Fogel EL, Easler JJ, Yuan Y, Yadav D, Conwell DL, Vege SS, Han SY, Park W, Patrick V, White FA. Safety, Tolerability, and Dose-Limiting Toxicity of Lacosamide in Patients With Painful Chronic Pancreatitis: Protocol for a Phase 1 Clinical Trial to Determine Safety and Identify Side Effects. JMIR Res Protoc. 2024 Mar 7;13:e50513. doi: 10.2196/50513. PMID 38451604